CLINICAL TRIAL: NCT07165457
Title: Clinical Evaluation of a Probiotic in Healthy Population (PROBIO)
Brief Title: Effect of Probiotic Intake in Healthy Population
Acronym: PROBIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PROBIO (2025.158)
Record Dates: First submitted 2025-08-12; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Adverse Effects; Healthy
Keywords: Probiotic; Supplement; Microbiota; Gastrointestinal tract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Probiotic group (Experimental): Capsule containing probiotic
  Interventions: Dietary Supplement: Probiotic group

INTERVENTIONS:
Dietary Supplement: Probiotic group — Daily consumption of one capsule containing a probiotic for 15 days

SUMMARY:
The main objective of this project is to evaluate the absence of adverse gastrointestinal effects following the consumption of a daily probiotic capsule during 15 days.

The secondary objective of this study is to verify the absence of any adverse effects other than gastrointestinal ones following the daily consumption of a probiotic during 15 days in a healthy population.

Specific objectives are:

* To evaluate changes in gastrointestinal health through self-reported questionnaire.
* To determine the adherence to probiotic consumption.
* To analyse headache, tiredness/fatigue, muscle or joint pain, fever or low-grade fever, chills, allergic reactions, difficulty sleeping, dizziness and general discomfort by General Adverse Effects Questionnaire.

Target sample size is 20 subjects.

Participants will be allocated in one group (experimental group).

Participants will visit nutritional intervention unit at Clinical Investigation Day 1 (day 1) and at Clinical Investigation Day 2 (day 15).

DETAILED DESCRIPTION:
Volunteers who wish to participate in the study will complete an online questionnaire to verify the main inclusion criteria. Those who meet the criteria will be invited to an information and screening visit to address any questions. Volunteers who agree to participate will sign the informed consent form.

During the intervention, participants will attend two clinical investigation visits. The first Clinical Investigation Day will be conducted on the same day as the screening, and the second Clinical Investigation Day will take place at the end of the 15-day period. In both visits, anthropometric measurements, gastrointestinal symptoms and a general questionnaire on adverse effects will be recorded. Volunteers will be required to consume one probiotic capsule per day during 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged between 18 and 70 years.
* Stable body weight (±5%) during the three months prior to study initiation.
* Physical examination and vital signs within normal limits or clinically irrelevant for the study.
* Subjects must be able to understand and willing to sign the informed consent form, and comply with all study procedures and requirements.
* Ongoing pharmacological/hormonal treatment will be permitted provided it does not affect the parameters under investigation and the dosage has been stable for at least three months prior to study initiation.
* Willingness to undergo all study procedures, including daily consumption of one probiotic capsule during the intervention.
* Availability in terms of time and location to attend the two scheduled in-person clinical evaluation sessions.

Exclusion Criteria:

* Volunteers undergoing pharmacological treatment with unstable dosing (less than 3 months prior to study initiation) will be excluded, particularly if treatments:
* Affect gastrointestinal function.
* Include chronically prescribed stomach protectants.
* Subjects with significant functional or structural abnormalities of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory or malabsorption diseases, hiatal hernia, chronic reflux, etc.
* Subjects who have undergone surgical procedures resulting in permanent alterations of the digestive system (e.g., gastroduodenostomy) or bariatric surgery.
* Presence of systemic intestinal, hepatic, or renal diseases, such as uncontrolled thyroid disorders, cirrhosis, inflammatory bowel disease, untreated anemia, etc. (non-alcoholic fatty liver disease will not be excluded).
* Alcohol consumption exceeding the sex-specific limits (>14 units/week for women, >20 units/week for men).
* Pregnancy, lactation, or plans to become pregnant during the study period.
* Use of nutritional supplements that may affect study outcomes (e.g., weight-loss supplements, newly initiated fiber supplements, probiotics, postbiotics, etc.).
* Subjects with any type of cancer currently undergoing treatment, or with less than five years since cancer remission.
* Known allergy to any component of the investigational product.
* Presence of cognitive and/or psychological impairments.
* Anticipated poor compliance or, in the investigator's opinion, difficulty adhering to study procedures.
* Participation in any weight loss or body composition modification treatments.
* Use of antibiotics within 15 days prior to the baseline visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-04 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-07 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Gastrointestinal symptoms will be registrated through Gastrointestinal Symptoms Rating Scale questionnaire, which is a questionnaire of 15 items. The questionnaire has a seven-point graded likert-type scale, where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.

SECONDARY OUTCOMES:
Body weight | Clinical Investigation Day 1
  Weight of participants will be measured by bioimpedance and reported in kg
Height | Clinical Investigation Day 1
  Height of participants will be measured by stadiometer and reported in m.
Body mass index | Clinical Investigation Day 1
  Body mass index will be calculated as follows: weight (kilograms)/ height (cm)2
Adherence to capsule consumption | Clinical Investigation Day 2
  Adherence will be assessed using the capsule consumption record form.
Headache | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Headache will be assess answering the General Questionnaire designed for the study. Answers could be None / Mild / Moderate / Severe.
Tiredness | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Tiredness will be assess answering the General Questionnaire designed for the study. Answers could be None / Mild / Moderate / Severe.
Muscle or joint pain | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Muscle or joint pain will be assess answering the General Questionnaire designed for the study. Answers could be None / Mild / Moderate / Severe.
Fever | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Fever will be assess answering the General Questionnaire designed for the study. Answers could be None / Mild / Moderate / Severe.
Chills | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Chills will be assess answering the General Questionnaire designed for the study. Answers could be None / Mild / Moderate / Severe.
Allergic reactions | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Allergic reactions will be assess answering the General Questionnaire designed for the study. Answers could be None / Mild / Moderate / Severe.
Difficulty sleeping | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Difficulty sleeping will be assess answering the General Questionnaire designed for the study. Answers could be None / Mild / Moderate / Severe.
Dizziness | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Dizziness will be assess answering the General Questionnaire designed for the study. Answers could be None / Mild / Moderate / Severe.
General discomfort | Clinical Investigation Day 1 and Clinical Investigation Day 2
  General discomfort will be assess answering the General Questionnaire designed for the study. Answers could be None / Mild / Moderate / Severe.
Mood | Clinical Investigation Day 2
  Mood will be assess answering the General Questionnaire designed for the study. Answers could be No / Yes, mild / Yes, moderate / Yes, severe
Other symptoms | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Open question

CONTACTS AND LOCATIONS:
Overall Officials: Idoia Ibero, PhD, Study Chair — Center for Nutrition Research; Salomé Pérez, Study Chair — Center for Nutrition Research; Paula Aranaz, PhD, Principal Investigator — Center for Nutrition Research; Verónica Ciaurriz, Study Chair — Center for Nutrition Research; Ana Lorente, Study Chair — Center for Nutrition Research
Locations (1):
- Center for Nutrition Research, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No